CLINICAL TRIAL: NCT02563379
Title: Association Between Circadian Blood Pressure Patterns With Asymptomatic Episodes of Paroxysmal Atrial Fibrillation in Hypertensive Subjects
Brief Title: Association of Dipping Pattern or Early Morning Surge of BP With Asymptomatic Episodes of Paroxysmal Atrial Fibrillation in Subjects With Hypertension (DIMOSPAF)
Acronym: DIMOSPAF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Emmanuel A. Andreadis, HEAD OF THE FOURTH INTERNAL MEDICINE DEPARTMENT, Evangelismos Hospital
Other Study IDs: MBPS-0915-EA
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension - Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Dippers: Dipping pattern is defined as daytime-nighttime BP/daytime BP reduction - based on either ABP monitoring- greater than 10% for systolic and/or diastolic BP.
  Extreme dipping is marked nocturnal systolic and/or diastolic BP fall>20% of daytime systolic and/or diastolic values or night/day systolic and/or diastolic BP ratio <0.8.
  Patients in this group will be dippers or extreme dippers. We aim to examine the association of this BP pattern with the development of asymptomatic episodes of paroxysmal atrial fibrillation, in hypertensive subjects.
- Non-dippers: Non-dipping and rising: no reduction or increase in nocturnal systolic and/or diastolic BP or night/day systolic and/or diastolic BP ratio ≥1.
  In this group we aim to examine whether an association exists between the non-dipping pattern and the development of asymptomatic episodes of paroxysmal atrial fibrillation in hypertensive subjects.
- Morning Hypertensives: It is known that morning surge is the excessive systolic and/or diastolic BP elevation rising in the morning.
  Patients in this group will have morning hypertension that is classified into two types:
  the "morning-surge" type, characterized by a marked increase in blood pressure in the early morning, and the "nocturnal-hypertension" type, characterized by high blood pressure that persists from nighttime until early morning.
  In our study we will examine whether an association between morning hypertension and asymptomatic episodes of paroxysmal atrial fibrillation exists in hypertensive subjects.

SUMMARY:
The goals of our study are to determine a).the association between abnormal circadian BP and the development of paroxysmal AF in hypertensive patients, b).at which level of TOD, paroxysmal AF episodes are detected in hypertensive subjects, c).if there is any association between systolic and/or diastolic BP levels with AF occurrence, d).whether the mean heart rate during a 24-hr interval is associated with the development of paroxysmal AF, and finally e).examine the relationship between a wide PP and asymptomatic AF episodes in patients with HTN.

DETAILED DESCRIPTION:
Atrial fibrillation, also known as AF or Afib, is an abnormal and irregular heart rhythm in which electrical signals are generated chaotically throughout the upper chambers (atria) of the heart. According to the NICE clinical guidelines, a patient who experiences recurrent (two or more) AF episodes that terminate spontaneously without any treatment in less than seven days, and usually within 48 hours is classified as having paroxysmal AF. It has been shown that paroxysmal AF comprises approximately between 25% and 62% of cases of AF, and it is estimated that both its incidence and prevalence are likely to rise as the worldwide population ages dramatically over the next twenty years. Interestingly, hospitalizations due to AF have increased sharply in the US during the last decade, posing thereby a heavy economic burden on the health care system and society.

Likewise, hypertension (HTN) also constitutes a major public health problem globally, and its prevalence is set to increase owing to widespread population ageing. This epidemiological trend is especially prevalent in rapidly developing countries where early routine screening at any point of health care is underutilized among risk subjects, due to several perceived barriers. Moreover, HTN awareness is critical for optimal BP control since under-diagnosis, under-treatment and/or un-treatment of high BP levels can have deleterious effects on the cardiovascular system. In addition, HTN is the single most important risk factor for cerebrovascular stroke, and it has been clearly demonstrated that it is also associated with structural and functional changes in the myocardium that favor the development of AF, further increasing the risk of thromboembolism. Among those alterations, left ventricular hypertrophy (LVH), impaired ventricular filling, left atrial enlargement and slowing of atrial conduction velocity have been identified as important heralds of cardiovascular morbidity and mortality. More specifically, since HTN and AF are two conditions that often co-exist, especially in patients with advanced age, the risk for considerable morbidity and mortality is increased even more, which points towards the significance that optimal BP control holds in the prevention of cardiovascular events. To our knowledge, in the Framingham Heart Study, after controlling for age and other predisposing conditions, HTN and diabetes emerged as the only cardiovascular risk factors predicting AF.

It has also been suggested that nocturnal HTN and non-dipping of BP during sleep are distinct entities that often occur together and are regarded as important harbingers of poor cardiovascular prognosis. Recently, Pierdomenico et al., showed that non-dipper sustained hypertensives have a two-fold greater risk of developing AF than dipper ones. This may be due to the fact that nighttime HTN may be a powerful determinant of long-standing left ventricular diastolic dysfunction, which subsequently increases atrial stretch. Furthermore, it has been observed that nighttime hemodynamics, are associated with higher sympathetic and reduced vagal activity, which may trigger AF. Additionally, sympathetic activation is associated with the stimulation of the renin-angiotensin-aldosterone axis (RAAA), which leads to increased left ventricular diastolic preload, both atrial and ventricular fibrosis, exerting thus direct cellular electrophysiological effects. Besides, scientists suggested that nighttime HTN is better associated with cardiovascular target organ damage (TOD) as compared with the non-dipping pattern.

According to the most recent guidelines of the ESH, the presence of microalbuminuria, increased pulse wave velocity, LVH on echocardiogram and carotid plaques detected during carotid ultrasonography, constitute markers of asymptomatic organ damage and it has been clearly demonstrated from multiple studies that they can predict CV mortality independently of SCORE stratification.

In our study we will try to investigate whether abnormalities in the circadian rhythm of BP (such as extreme dipping or non-dipping pattern, and/or morning surge) in hypertensive subjects with or without TOD are associated with the development of new-onset paroxysmal AF.

24-hr ambulatory BP monitoring (ABPM) along with the 24-hour blood pressure monitors with AF detector will help us to examine the incidence of AF in extremely dippers or non-dippers, and/or patients exhibiting a morning surge in BP, with or without TOD. Some of the questions that we aim to answer while conducting this study are whether an asymptomatic AF episode is more commonly detected in extreme dippers, non-dippers, or morning surgers, during daytime or during nighttime, or whether TOD is associated with asymptomatic AF episodes.

Importantly, Iqbal et al, demonstrated that there is an association between AF and nighttime DBP. On top of that, during the past decade, a research study conducted in 546 hypertensive subjects aged < 60 years of age and who were followed-up for 9.2 years, showed that DBP, whether 24-hr mean, daytime mean, or nighttime mean, provided the most incremental value for the prediction of morbid events. Thereby, we want to examine if AF episodes have any association with the 24hr systolic and the diastolic blood pressure (DBP) levels. It would also be interesting to observe for any associations between AF occurrence and the mean 24-hr ABPM and office heart rate (HR).

Moreover, it has been showed that pulse pressure (PP) determines left atrial enlargement in non-dipper patients with never-treated essential HTN. Thus, in our study, we will also examine whether a wide PP is associated with silent AF episodes in treated hypertensive subjects.

Summarizing, the goals of our study are to determine a).the association between abnormal circadian BP and the development of paroxysmal AF in hypertensive patients, b).at which level of TOD, paroxysmal AF episodes are detected in hypertensive subjects, c).if there is any association between systolic and/or diastolic BP levels with AF occurrence, d).whether the mean heart rate during a 24-hr interval is associated with the development of paroxysmal AF, and finally e).examine the relationship between a wide PP and asymptomatic AF episodes in patients with HTN.

Study Population We will evaluate all adult patients referred by their family physicians to the "Hypertension and Cardiovascular Prevention" Outpatient Clinic at Evangelismos General Hospital in Athens, from June 2015 to present.

All patients with an average office systolic BP ≥140 mmHg and/or an average diastolic BP ≥90 mmHg on three consecutive visits are considered as having essential HTN. Furthermore, individuals under treatment with one or more antihypertensive drug are also enrolled in the study.

Objectives Primary endpoint

• To investigate whether nighttime BP patterns (extreme dipping, normal dipping or reduced dipping and non-dipping including risers) or early morning surge are associated with the detection of paroxysmal AF in hypertensive subjects.

Further definitions Normal diurnal systolic and diastolic BP pattern: arterial BP has a daily variation characterized by substantial reductions during sleep, a rapid rise upon awakening, and increased variability during the awake period in ambulant normal subjects and hypertensive patients.

Reduced diurnal systolic and diastolic BP pattern: nocturnal systolic and/or DBP fall from 1 to 10% of daytime values or night/day systolic and/or diastolic BP ratio <1 and >0.9.

Nocturnal HTN: increased absolute level of night time systolic and/or diastolic BP (≥120/70 mmHg).19 Dipping pattern is defined as daytime-nighttime BP/daytime BP reduction - based on either ABP or home BP (HBP) monitoring- greater than 10% for systolic and/or diastolic BP. Nighttime HTN is defined as nighttime ABP or HBP ≥125/75 mmHg (systolic and/or diastolic).

Non-dipping and rising: no reduction or increase in nocturnal systolic and/or diastolic BP or night/day systolic and/or diastolic BP ratio ≥1.

Extreme dipping: marked nocturnal systolic and/or diastolic BP fall>20% of daytime systolic and/or diastolic values or night/day systolic and/or diastolic BP ratio <0.8.

Morning surge: excessive systolic and/or diastolic BP elevation rising in the morning.

Secondary endpoints

* To detect asymptomatic and intermittent AF using a 24h ABPM with atrial fibrillation detector device and to compare its accuracy with Holter monitoring.
* To investigate the agreement in the detection of paroxysmal AF using simultaneously the 24h-ABP with AF detection device and loop recording.
* To observe at which level of TOD, asymptomatic AF episodes are more commonly detected.
* To study if there is any relationship between systolic and/or diastolic BP levels with AF occurrence.
* To examine whether office HR or mean HR using ABPM is associated with the development of silent AF episodes.
* To examine whether a wide PP in ABPM is associated with the development of silent AF episodes.

Variables used to determine the primary and secondary endpoints

* Sociodemographic data (birth date, gender, education level, employment status, place of residence, smoking status/habits, alcohol consumption)
* Anthropometric characteristics (body weight, height, waist circumference)
* Any abnormal findings on physical examination
* Clinical relevant medical history and comorbidities
* Concomitant medications
* Electrocardiographic assessment
* Investigation of TOD, including echocardiography, carotid artery triplex, 24h-urine albumin excretion and ABI
* Recent laboratory testing results including hemoglobin, hematocrit, blood glucose, kidney and liver function tests
* Management of HTN (pharmacologic and non-pharmacologic treatment)

Inclusion Criteria

* Patients diagnosed with essential HTN (office BP>140/90mmHg) or patients receiving at least one antihypertensive medication (ie. RAAA inhibitors or diuretic), aged 18-85 years of age.
* Patients with at least one of the following risk factors, organ damage or other evidence of cardiovascular disease:
* Previous stroke
* Transient ischemic attack (TIA)
* Systemic embolism
* Diabetes mellitus type 2
* Obesity
* Obstructive sleep apnea (OSA)
* Dyslipidemia
* History of coronary artery disease (CAD)
* Valvular heart disease (VHD)
* Echocardiographic findings attributed to HTN (ie. diastolic dysfunction, LVH)
* White coat hypertension (WCH), masked hypertension (MH)
* Positive family history for rhythm disturbances

Exclusion Criteria

* Patients already diagnosed with paroxysmal or permanent AF
* Severe renal insufficiency (eGFR according to MDRD formula <25ml/min/1.73m2)
* Patients unable to attend follow-up visits
* Clinical evidence of severe heart failure
* Suspected secondary HTN
* Mental disorders
* Patients with cancer

The study protocol needs to be approved by the scientific board of the hospital and signed informed consent needs to be obtained from all participants.

Study Design We are going to conduct a cross-sectional, observational study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with essential HTN (office BP>140/90mmHg) or patients receiving at least one antihypertensive medication (ie. RAAA inhibitors or diuretic), aged 18-85 years of age.
* Patients with at least one of the following risk factors, organ damage or other evidence of cardiovascular disease:
* Previous stroke
* Transient ischemic attack (TIA)
* Systemic embolism
* Diabetes mellitus type 2
* Obesity
* Obstructive sleep apnea (OSA)
* Dyslipidemia
* History of coronary artery disease (CAD)
* Valvular heart disease (VHD)
* Echocardiographic findings attributed to HTN (ie. diastolic dysfunction, LVH)
* White coat hypertension (WCH), masked hypertension (MH)
* Positive family history for rhythm disturbances

Exclusion Criteria:

* Patients already diagnosed with paroxysmal or permanent AF
* Severe renal insufficiency (eGFR according to MDRD formula <25ml/min/1.73m2)
* Patients unable to attend follow-up visits
* Clinical evidence of severe heart failure
* Suspected secondary HTN
* Mental disorders
* Patients with cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will evaluate all adult patients referred by their family physicians to the "Hypertension and Cardiovascular Prevention" Outpatient Clinic at Evangelismos General Hospital in Athens, from June 2015 to present.
  All patients with an average office systolic BP ≥140 mmHg and/or an average diastolic BP ≥90 mmHg on three consecutive visits are considered as having essential HTN. Furthermore, individuals under treatment with one or more antihypertensive drug are also enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Association between nighttime BP patterns and/or early morning surge with the development of asymptomatic episodes of paroxysmal atrial fibrillation in hypertensive subjects | 12 months
  • To investigate whether nighttime BP patterns (extreme dipping, normal dipping or reduced dipping and non-dipping including risers) or early morning surge are associated with the detection of paroxysmal AF in hypertensive subjects.

SECONDARY OUTCOMES:
Association between the degree of TOD and the development of paroxysmal AF in hypertensive patients | 12 months
  • To observe at which level of TOD, asymptomatic AF episodes are more commonly detected.
Association between SBP and/or DBP levels with the development of paroxysmal AF in hypertensive patients | 12 months
  • To study if there is any relationship between systolic and/or diastolic BP levels with AF occurrence.
Association between office heart rate or mean 24-hr heart rate with the development of asymptomatic paroxysmal AF episodes. | 12 months
  • To examine whether office HR or mean HR using ABPM is associated with the development of silent AF episodes.
Association between PP and the development of asymptomatic paroxysmal AF episodes | 12 months
  • To examine whether a wide PP in ABPM is associated with the development of silent AF episodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelismos General Hospital, Athens, Attica, Greece

REFERENCES:
- [Result] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D. 2012 HRS/EHRA/ECAS Expert Consensus Statement on Catheter and Surgical Ablation of Atrial Fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design. Europace. 2012 Apr;14(4):528-606. doi: 10.1093/europace/eus027. Epub 2012 Mar 1. No abstract available. PMID 22389422
- [Result] Lip GY, Hee FL. Paroxysmal atrial fibrillation. QJM. 2001 Dec;94(12):665-78. doi: 10.1093/qjmed/94.12.665. PMID 11744787
- [Result] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Result] Patel NJ, Deshmukh A, Pant S, Singh V, Patel N, Arora S, Shah N, Chothani A, Savani GT, Mehta K, Parikh V, Rathod A, Badheka AO, Lafferty J, Kowalski M, Mehta JL, Mitrani RD, Viles-Gonzalez JF, Paydak H. Contemporary trends of hospitalization for atrial fibrillation in the United States, 2000 through 2010: implications for healthcare planning. Circulation. 2014 Jun 10;129(23):2371-9. doi: 10.1161/CIRCULATIONAHA.114.008201. Epub 2014 May 19. PMID 24842943
- [Result] Tibazarwa KB, Damasceno AA. Hypertension in developing countries. Can J Cardiol. 2014 May;30(5):527-33. doi: 10.1016/j.cjca.2014.02.020. Epub 2014 Mar 4. PMID 24786443
- [Result] Sarafidis PA, Li S, Chen SC, Collins AJ, Brown WW, Klag MJ, Bakris GL. Hypertension awareness, treatment, and control in chronic kidney disease. Am J Med. 2008 Apr;121(4):332-40. doi: 10.1016/j.amjmed.2007.11.025. PMID 18374693
- [Result] Rundek T, Sacco RL. Risk factor management to prevent first stroke. Neurol Clin. 2008 Nov;26(4):1007-45, ix. doi: 10.1016/j.ncl.2008.09.001. PMID 19026901
- [Result] Healey JS, Connolly SJ. Atrial fibrillation: hypertension as a causative agent, risk factor for complications, and potential therapeutic target. Am J Cardiol. 2003 May 22;91(10A):9G-14G. doi: 10.1016/s0002-9149(03)00227-3. PMID 12781903
- [Result] Kannel WB, Wolf PA, Benjamin EJ, Levy D. Prevalence, incidence, prognosis, and predisposing conditions for atrial fibrillation: population-based estimates. Am J Cardiol. 1998 Oct 16;82(8A):2N-9N. doi: 10.1016/s0002-9149(98)00583-9. PMID 9809895
- [Result] de la Sierra A, Gorostidi M, Banegas JR, Segura J, de la Cruz JJ, Ruilope LM. Nocturnal hypertension or nondipping: which is better associated with the cardiovascular risk profile? Am J Hypertens. 2014 May;27(5):680-7. doi: 10.1093/ajh/hpt175. Epub 2013 Sep 23. PMID 24061070
- [Result] Pierdomenico SD, Lapenna D, Cuccurullo F. Risk of atrial fibrillation in dipper and nondipper sustained hypertensive patients. Blood Press Monit. 2008 Aug;13(4):193-7. doi: 10.1097/MBP.0b013e3282feea70. PMID 18635973
- [Result] Tsioufis C, Andrikou I, Thomopoulos C, Syrseloudis D, Stergiou G, Stefanadis C. Increased nighttime blood pressure or nondipping profile for prediction of cardiovascular outcomes. J Hum Hypertens. 2011 May;25(5):281-93. doi: 10.1038/jhh.2010.113. Epub 2010 Dec 2. PMID 21124340
- [Result] Iqbal P, Stevenson L. Cardiovascular outcomes in patients with normal and abnormal 24-hour ambulatory blood pressure monitoring. Int J Hypertens. 2010 Dec 5;2011:786912. doi: 10.4061/2011/786912. PMID 21151547
- [Result] Khattar RS, Swales JD, Dore C, Senior R, Lahiri A. Effect of aging on the prognostic significance of ambulatory systolic, diastolic, and pulse pressure in essential hypertension. Circulation. 2001 Aug 14;104(7):783-9. doi: 10.1161/hc3201.094227. PMID 11502703
- [Result] Triantafyllidi H, Ikonomidis I, Lekakis J, Panou F, Georgoula G, Fountoulaki K, Kremastinos D. Pulse pressure determines left atrial enlargement in non-dipper patients with never-treated essential hypertension. J Hum Hypertens. 2007 Nov;21(11):897-9. doi: 10.1038/sj.jhh.1002236. Epub 2007 May 31. No abstract available. PMID 17541387
- [Result] Deyneli O, Yazici D, Toprak A, Yuksel M, Aydin H, Tezcan H, Yavuz DG, Akalin S. Diurnal blood pressure abnormalities are related to endothelial dysfunction in patients with non-complicated type 1 diabetes. Hypertens Res. 2008 Nov;31(11):2065-73. doi: 10.1291/hypres.31.2065. PMID 19098379
- [Result] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ; Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Recommendations for blood pressure measurement in humans and experimental animals: Part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Hypertension. 2005 Jan;45(1):142-61. doi: 10.1161/01.HYP.0000150859.47929.8e. Epub 2004 Dec 20. PMID 15611362
- [Result] Millar-Craig MW, Bishop CN, Raftery EB. Circadian variation of blood-pressure. Lancet. 1978 Apr 15;1(8068):795-7. doi: 10.1016/s0140-6736(78)92998-7. PMID 85815
- [Result] Parati G, Stergiou G, O'Brien E, Asmar R, Beilin L, Bilo G, Clement D, de la Sierra A, de Leeuw P, Dolan E, Fagard R, Graves J, Head GA, Imai Y, Kario K, Lurbe E, Mallion JM, Mancia G, Mengden T, Myers M, Ogedegbe G, Ohkubo T, Omboni S, Palatini P, Redon J, Ruilope LM, Shennan A, Staessen JA, vanMontfrans G, Verdecchia P, Waeber B, Wang J, Zanchetti A, Zhang Y; European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. European Society of Hypertension practice guidelines for ambulatory blood pressure monitoring. J Hypertens. 2014 Jul;32(7):1359-66. doi: 10.1097/HJH.0000000000000221. PMID 24886823
- [Result] Verdecchia P, Angeli F, Mazzotta G, Garofoli M, Ramundo E, Gentile G, Ambrosio G, Reboldi G. Day-night dip and early-morning surge in blood pressure in hypertension: prognostic implications. Hypertension. 2012 Jul;60(1):34-42. doi: 10.1161/HYPERTENSIONAHA.112.191858. Epub 2012 May 14. PMID 22585951